CLINICAL TRIAL: NCT05952635
Title: Tip Bendable Suction Ureteral Access Sheath vs. Traditional Ureteral Access Sheath in Retrograde Intrarenal Stone Surgery (RIRS): Study Protocol of a Multicentre, Prospective, Single-blinded, Randomized Controlled Trial
Brief Title: Tip Bendable Suction Ureteral Access Sheath vs. Traditional Ureteral Access Sheath in Retrograde Intrarenal Stone Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Xiangya Hospital of Central South University (Other); Xinchang County Hospital of Traditional Chinese Medicine (Unknown); Prof. Dr. Ilhan Varank Education and Training Hospital (Unknown); Jose R. Reyes Memorial Medical Center (Other Government); Guizhou Provincial People's Hospital (Other); University of Malaya (Other)
Responsible Party: Principal Investigator, Guohua Zeng, Vice president, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MRER2023-001
Record Dates: First submitted 2023-06-17; First posted 2023-07-19 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Kidney Stone
Keywords: Kidney stone; Flexible ureteroscopy; Ureteral access sheath
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tip bendable suction ureteral access sheath (S-UAS) group (Experimental): Patients will use S-UAS during flexible ureteroscopy.
  Interventions: Procedure: Tip bendable suction ureteral access sheath
- Traditional ureteral access sheath group (No Intervention): Patients will use traditional UAS during flexible ureteroscopy.

INTERVENTIONS:
Procedure: Tip bendable suction ureteral access sheath — Patient use tip bendable suction ureteral access sheath during flexible ureteroscopy to see if flexible ureteroscopy with S-UAS offers the better treatment outcomes in terms of clinical effectiveness and post-operative complications.
  Arms: Tip bendable suction ureteral access sheath (S-UAS) group

SUMMARY:
Nephrolithiasis is the most common chronic kidney condition and affecting approximately one in every 10-17 people in the world[1,2]. Flexible ureteroscopy (f-URS) has become one of the most common treatments for ureteral and renal stones with minimal complications. The development of ureteral access sheath (UAS) is a significant advance in flexible ureteroscopic management of urinary stones. The UAS has two major advantages: 1) facilitating multiple entries into the renal collecting system without causing recurrent trauma to the ureter and permit expeditious basketing of multiple stone fragments, 2) improving the irrigation with better fluid outflow, thereby reducing the renal pelvic pressure (RPP) and risk of infectious complications.

The tip bendable suction ureteral access sheath (S-UAS) is a novel UAS that has good flexibility and deformability at the tip, which can passively bend (bend >90°) with the bending of f-URS and can connect to a vacuum suction device. Preliminary study showed that S-UAS can follow f-URS to cross the UPJ and into the renal pelvis and calices. S-UAS close to the stone can achieve complete stone-free status in RIRS. However, further clinical studies and comparisons with available techniques are required. This prospective, single-blinded, single-center, randomized control trial will evaluate the stone free rates, operative time, postoperative complications following RIRS with S-UAS. To the best of our knowledge, this is the first study to compare the clinical benefits of RIRS with S-UAS and traditional UAS.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ 18 years;
* American Society of Anesthesiology score 1-3;
* Upper urinary stone (kidney stone or upper ureteral stone) diameter of ≤ 3 cm confirmed by CT;
* Capable of giving written informed consent, which includes adherence with the requirements of the trial.

Exclusion Criteria:

* Patients with abnormal urinary tract anatomy (such as horseshoe kidney or ileal conduit);
* Patients with uncontrolled UTI;
* Patients with health or other factors that are absolute contraindications to RIRS;
* Patients unable to understand or complete trial documentation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2023-08-02 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
Immediate stone-free rate | Postoperative day 1
  No residual stone, or no stone fragments larger than 2 mm on KUB and ultrasound at postoperative day 1 are defined as stone free.

SECONDARY OUTCOMES:
Stone-free rate at 3 months | Postoperative 3 month
  No residual stone, or no stone fragments larger than 2 mm on CT scan at postoperative 3 month are defined as stone free.
Duration of hospital stay | From date of operation until the date of discharge, assessed up to 2 weeks.
Further interventions received up to 3 months post randomization | Postoperative 3 month
Complications up to 3 months post randomization | Postoperative 3 month
Change of Quality of life Score (prior to surgery and at month 3 after randomization) | Postoperative 3 month
Operative time | From start of operation until the end of operation, assessed up to 2 weeks.
  The duration from the insertion of the endoscope into the urethra to the completion of stent placement.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhu W, Liu S, Cao J, Wang H, Liang H, Jiang K, Cui Y, Chai CA, Sahinler EB, Aquino A, Mazzon G, Zhong W, Zhao Z, Zhang L, Ding J, Wang Q, Wang Y, Chen KW, Liu Y, Choong S, Sarica K, Zeng G. Tip bendable suction ureteral access sheath versus traditional sheath in retrograde intrarenal stone surgery: an international multicentre, randomized, parallel group, superiority study. EClinicalMedicine. 2024 Jul 5;74:102724. doi: 10.1016/j.eclinm.2024.102724. eCollection 2024 Aug. PMID 39070176